CLINICAL TRIAL: NCT00736762
Title: Effects of Global Postural re-Education Program on the Biomechanical Characteristics of the Elderly Balance.
Brief Title: Effects of Global Postural re-Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Gilmar Moraes Santos / PhD, University of the State of Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 136/07
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-08

CONDITIONS: Healthy; Elderly
Keywords: Global postural re-education; Balance; Physical therapy; older people

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- GPR (Experimental): Global postural re-education intervention
  Interventions: Other: GPR

INTERVENTIONS:
Other: GPR — The subjects randomised to the GPR program will participate in posture retraining techniques of approximately forty minutes, one time a week for ten weeks.

SUMMARY:
The postural alterations present in the seniors people act as predisponent form of incapacities that provoke alterations in the quality of life. The objective of this study is to evaluate the biomechanical characteristics of the balance of elderly people, before and after treatment with Global Postural Re-education. This research is characterized by experimental method of investigation.Thirty elderly people (30 women) will be randomized to two different groups from Group of Studies of Third Age - GETI, at University of the State of Santa Catarina:

* fifteen elderly women will be submitted to the Global Postural Re-education (GPR) program and to the GETI program of activities
* fifteen elderly women will be submitted only to the GETI program of activities.

At baseline the subjects will be screened for balance measurements with the chattecx balance system and Berg Scale. These measurements will be repeat immediately after the intervention. The subjects randomised to the GPR program will participate in posture retraining techniques of approximately forty minutes, one time a week for ten weeks. The independent t test for pairs of random samples will be used, with level of significance of p≤0,05.

ELIGIBILITY:
Inclusion Criteria:

* Senior that accomplish physical activity in the GETI (group of studies of the third age - Santa Catarina State University)

Exclusion Criteria:

* Visually impaired person
* Vestibular disorder
* Neurologic disorders
* Use of prostheses and ortheses
* Cancer

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2008-04 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
center of pressure (cop) | pre-treatment, five weeks and pos-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gilmar Santos, PhD, Principal Investigator — Santa Catarina State University
Locations (1):
- Santa Catarina State University, Florianópolis, Santa Catarina, Brazil